CLINICAL TRIAL: NCT04483323
Title: Erector Spinae Plane Block Versus Intraarticular Injection of Local Anesthetic for Postoperative Analgesia in Patients Undergoing Shoulder Arthroscopy; A Prospective Randomized Controlled Study
Brief Title: Erector Spinae Plane Block Versus Intraarticular Injection for Postoperative Analgesia in Shoulder Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Taysser Mahmoud Abdalraheem, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 33097/04/19
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Shoulder Arthroscopy; Postoperative Analgesia; Erector Spinae Plane Block; Intraarticular Injection
MeSH Terms: interventions — Injections, Intra-Articular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: Intraarticular group ( IA ) (Active Comparator): Patients will receive 20 ml of 0.25% bupivacaine intra-articularly through the surgical port
  Interventions: Procedure: Intraarticular Injection
- Group II: Erector Spinae Plane Block group ( ES ) (Experimental): Patients will receive an ultrasound guided erector spinae plane block using 20 ml of 0.25% bupivacaine at the level of T2 transverse process
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — The patient will be placed in the lateral position. Following skin disinfection, counting down from the C7 spinous process and using ultrasound guidance, the level of T2 transverse process will be identified. A 2-5 MH2 curved array transducer (sono site Edge, Bothell, Will behington) will be positioned transversely to visualize the lateral tip of T2 transverse Process. A longitudinal parasagittal orientation will be obtained over the transverse process using a 22 - gauge 8 cm block needle (visioplex, Vygon , France) will be inserted in plane to US beam in a caudal to cranial direction to place the needle tip between the posterior fascia of the erector spinae muscle and the T2 transverse process.
  Position of the needle tip in the ESP deep to the erector spinae muscle will be confirmed using hydrodissection with 0.5 - 1 ml of normal saline and visualization of the linear fluid spread deep to the erector spinae muscle following which 20 ml of 0.25% bupivacaine will be injected.
  Arms: Group II: Erector Spinae Plane Block group ( ES )
Procedure: Intraarticular Injection — Intraarticular injection of local anesthetic through the surgical port
  Arms: Group I: Intraarticular group ( IA )

SUMMARY:
To improve the outcome after surgery, effective pain control is needed. The aim of the current study was to compare the efficacy of ultrasound guided erector spinae plane block versus the intra articular injection of local anesthetic for post-operative analgesia in patients undergoing shoulder arthroscopy.

DETAILED DESCRIPTION:
Sample size calculation:

Calculation of sample size was done to detect a 15% difference in the VAS score between two groups detected that at least 27 patients were needed at an α error of 0.05 and 80 % power of the study. The number will be increased to 30 patients to avoid a 10% dropped out patients.

Statistical analysis Statistical analysis will be done by Statistical Package for the Social Sciences (SPSS) v25 (IBM Inc., Chicago, USA). Normality of data will be checked with Shapiro-Wilks test and histogram. Quantitative variables will be presented as mean and standard deviation (SD) and will be compared by unpaired student T test. Categorical variables will be presented as frequency and percentage (%) and will be analysed by the Chi-square test. P value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-II
* Posted for elective shoulder arthroscopy

Exclusion Criteria:

* Coagulopathy
* Allergy to local anesthetics
* Chronic use of narcotics
* Necessity for an intra articular drain after surgery
* Patients refusal to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
The amount of total postoperative rescue analgesic consumption (mg) | First 24 hours postoperative
  Rescue analgesia in the form of diclofenac sodium 75mg intramuscularly (IM) will be given if the visual analogue scale ≥ 40

SECONDARY OUTCOMES:
Postoperative visual analogue scale | First 24 hours postoperative
  Visual analogue scale (VAS) for determination of intensity of the pain on scale from (0-100) where 0= no pain and 100=the worst pain.

OTHER OUTCOMES:
The time to first request of rescue analgesia (hours) | First 24 hours postoperative
  Time till the first need of rescue analgesia in the form of diclofenac sodium 75mg postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Taysser M Abdelraheem, MD, Principal Investigator — Lecturer at Tanta University Hospitals
Locations (1):
- Tanta University Hospitals, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: No